CLINICAL TRIAL: NCT03890172
Title: Efficacy of Platelets Rich Plasma as a Therapeutic Tool in Chronic Non Healing Diabetic Foot Ulcers
Brief Title: Efficacy of Platelets Rich Plasma as a Therapeutic Tool in Diabetic Foot Ulcers
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hanaa Mohammed Riad, assistant lecture, Assiut University
Other Study IDs: Platelets rich plasma
Record Dates: First submitted 2019-03-15; First posted 2019-03-26 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Diabetic Foot Ulcer
Keywords: platelets rich plasma
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study group: in this group the investigators will be managing diabetic wounds with platelet rich plasma treatment.
  Interventions: Other: 20-100 ml venous blood will be drawn the from patient into sterilized centrifuge tube ,following centrifuge to separate PRP and at the bed side and tricked onto the ulcer twice weekly
- control group: In this group patients will receive the standard treatment in form of debridement and dressing twice weekly
  Interventions: Other: standard treatment

INTERVENTIONS:
Other: 20-100 ml venous blood will be drawn the from patient into sterilized centrifuge tube ,following centrifuge to separate PRP and at the bed side and tricked onto the ulcer twice weekly — topical application of platelets rich plasma after Centrifugation at diabetic foot ulcer to study group ,history taking . Ankle brachial index (ABI) measuring and laboratory testes including hemoglobin A1c ( HgA1)c,cbc and prothrombin time( pt) and prothrombin concentration ( pc)
  Groups: study group
Other: standard treatment — Subjects in the control group will receive Standard Wound Care treatment for chronic ulcers according to accepted medical practices.
  Groups: control group

SUMMARY:
using platelet-rich plasma (PRP) in healing diabetic foot ulcers (DFUs), and to compare the rate of healing and final outcome with conventional therapy.

DETAILED DESCRIPTION:
Diabetic foot ulcers (DFU) are one of the most frequent and difficult complications in diabetes. The risk for a diabetic patient to develop an ulcer during his life is estimated as being 25%. Ulcers are a frequent cause of lower limbs amputation and 84% of lower limb amputations are preceded by ulcers .

Diabetic ulcer (DU) is not only a serious clinical problem with negative impacts on both the life quality and survival time, but also an economic burden with significant contribution to high cost and lengthy hospitalizations. Furthermore, the non healing diabetic cutaneous ulcers along with the subsequent amputations may bring about costly to treat and painful disabilities. However, healing of the DU may be improved and most of the amputations may be prevented by more effective treatments based on diabetic education .

In spite of the high prevalence and morbidity associated with DFUs, current treatment options are limited. Current standard management consists of surgical debridement followed by frequent dressing changes with tight infection and glycemic control. Despite this comprehensive approach, complication and amputation rates remain high.

The use of platelet-rich plasma (PRP) has emerged as an adjunctive method for treating DFUs.

Platelet-rich plasma (PRP) preparations were first described in the 1980s as plasma with a platelet count above that found normally in peripheral blood.

First used in the field of hematology, PRP use has expanded throughout the fields of dermatology, oral-maxillofacial surgery, plastic surgery, cardiac surgery, ophthalmology, urology, and gynecology .

The concentration of platelets in PRP is 2-6 folds higher than that of whole blood .

The curative properties of PRP rely on the fact that platelets are a physiological reservoir of a variety of growth factors, with healing function which have an active role in tissue regeneration .

Platelets contain proteins, known as growth factors that trigger biological effects including directed cell migration (i.e. chemotaxis), angiogenesis, cell proliferation and differentiation, which are key elements in the process of tissue repair and regeneration.

Specifically, the platelet alpha-granules contain several of these molecules, including: platelet derived growth factor (PDGF),transforming growth factor B ( TGF-β), vascular endothelial growth factor (VEGF), epithelial growth factor (EGF), fibrinogen, fibronectin, and vitronectin.

In addition, platelet delta granules contain serotonin, histamine, dopamine, calcium, and adenosine, which act in tandem with the aforementioned growth factors to regulate wound healing .

platelets exert antimicrobial activity against some bacteria of the skin, and clinical data shows that the presence of infection is reduced in PRP-treated wounds.

The advantages and merits of PRP are apparent since it is easy, cost-effective and much more lasting compared to other standard treatments and being autologous in nature, it is free from communicable pathogens, making it a safe treatment modality with good clinical results

ELIGIBILITY:
Inclusion Criteria:

* diabetic patients 18 to 80 years of age, with at least one cutaneous ulcer, which did not improve significantly after at least 4 week ulcer standard treatments
* ankle brachial index value ≥ 0.6
* platelet count ≥ 100,000 /mm 3
* no history of various drug or dressing allergies

Exclusion Criteria:

* - ulcer is due to non diabetic etiology
* patients blood vessels are non compressible for ankle brachial index (ABI )testing
* the presence of an infected wound and/or osteomyelitis, and/or a completely necrotic ulcer
* active oncological disease. systemic treatment medications like corticosteroids, immunosuppressive agents, as well as radiation or chemotherapy at the target sites within 3 weeks before this study.
* Screening platelets count less than 100,000mm3
* Screening hemoglobin less than10.5mg/dl
* End stages renal disease,haematological,collagen vascular disease and bleeding disorders

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: , The study included 60 patients of both sex from 18 to 80 years, with clean chronic diabetic foot ulcers divided into 2 equal groups. The study group in which PRP was used, and the control group receiving standard therapy The formed PRP was applied to the wound twice weekly.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-07-30 (Estimated); Primary Completion 2021-10-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Change of ulcer size | 16 weeks
  ulcer size will be measured with ruler/probe for length, width and depth and estimated by calculating the ulcer size in centimeter (cm 2).

SECONDARY OUTCOMES:
time of wound healing | 16 weeks
  Complete wound closure over period of 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hanan Mohamoud, Study Director — Assiut University
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bernuzzi G, Tardito S, Bussolati O, Adorni D, Cantarelli S, Fagnoni F, Rossetti A, Azzarone M, Ficarelli E, Caleffi E, Gazzola G, Franchini M. Platelet gel in the treatment of cutaneous ulcers: the experience of the Immunohaematology and Transfusion Centre of Parma. Blood Transfus. 2010 Oct;8(4):237-47. doi: 10.2450/2009.0118-09. PMID 20967164
- [Background] Piccin A, Di Pierro AM, Canzian L, Primerano M, Corvetta D, Negri G, Mazzoleni G, Gastl G, Steurer M, Gentilini I, Eisendle K, Fontanella F. Platelet gel: a new therapeutic tool with great potential. Blood Transfus. 2017 Jul;15(4):333-340. doi: 10.2450/2016.0038-16. Epub 2016 Jul 25. PMID 27483482
- [Background] Apelqvist J, Bakker K, van Houtum WH, Schaper NC; International Working Group on the Diabetic Foot (IWGDF) Editorial Board. The development of global consensus guidelines on the management of the diabetic foot. Diabetes Metab Res Rev. 2008 May-Jun;24 Suppl 1:S116-8. doi: 10.1002/dmrr.832. PMID 18442162
- [Background] Everett E, Mathioudakis N. Update on management of diabetic foot ulcers. Ann N Y Acad Sci. 2018 Jan;1411(1):153-165. doi: 10.1111/nyas.13569. PMID 29377202
- [Background] Mohammadi MH, Molavi B, Mohammadi S, Nikbakht M, Mohammadi AM, Mostafaei S, Norooznezhad AH, Ghorbani Abdegah A, Ghavamzadeh A. Evaluation of wound healing in diabetic foot ulcer using platelet-rich plasma gel: A single-arm clinical trial. Transfus Apher Sci. 2017 Apr;56(2):160-164. doi: 10.1016/j.transci.2016.10.020. Epub 2016 Nov 2. PMID 27839965
- [Background] Alves R, Grimalt R. A Review of Platelet-Rich Plasma: History, Biology, Mechanism of Action, and Classification. Skin Appendage Disord. 2018 Jan;4(1):18-24. doi: 10.1159/000477353. Epub 2017 Jul 6. PMID 29457008
- [Background] Andia E R-AJ, Martin I, Abate M. Current concepts and translational uses of platelet rich plasma biotechnology. Biotechnology 2015. https://doi.org/10.5772/59954 Google Scholar
- [Background] San Sebastian KM, Lobato I, Hernandez I, Burgos-Alonso N, Gomez-Fernandez MC, Lopez JL, Rodriguez B, March AG, Grandes G, Andia I. Efficacy and safety of autologous platelet rich plasma for the treatment of vascular ulcers in primary care: Phase III study. BMC Fam Pract. 2014 Dec 30;15:211. doi: 10.1186/s12875-014-0211-8. PMID 25547983
- [Background] Andia I, Abate M. Platelet-rich plasma: underlying biology and clinical correlates. Regen Med. 2013 Sep;8(5):645-58. doi: 10.2217/rme.13.59. PMID 23998756
- [Background] Anitua E, Aguirre JJ, Algorta J, Ayerdi E, Cabezas AI, Orive G, Andia I. Effectiveness of autologous preparation rich in growth factors for the treatment of chronic cutaneous ulcers. J Biomed Mater Res B Appl Biomater. 2008 Feb;84(2):415-21. doi: 10.1002/jbm.b.30886. PMID 17595032
- [Background] Kakudo N, Kushida S, Ogura N, Hara T, Suzuki K. The use of autologous platelet rich plasma in the treatment of intractable skin ulcer. Open J Reg Med. 2012;1:29-32. N, Kushida S, Ogura N, Hara T, Suzuki K. The use of autologous platelet rich plasma in the treatment of intractable skin ulcer. Open J Reg Med. 2012;1:29-32.
- [Background] Liao HT, Marra KG, Rubin JP. Application of platelet-rich plasma and platelet-rich fibrin in fat grafting: basic science and literature review. Tissue Eng Part B Rev. 2014 Aug;20(4):267-76. doi: 10.1089/ten.TEB.2013.0317. Epub 2013 Dec 18. PMID 24004354
- [Background] Carter MJ, Fylling CP, Parnell LK. Use of platelet rich plasma gel on wound healing: a systematic review and meta-analysis. Eplasty. 2011;11:e38. Epub 2011 Sep 15. PMID 22028946
- [Background] Lacci KM, Dardik A. Platelet-rich plasma: support for its use in wound healing. Yale J Biol Med. 2010 Mar;83(1):1-9. PMID 20351977